CLINICAL TRIAL: NCT02029053
Title: VR101: A Pilot Study to Evaluate the Preliminary Feasibility and Safety of a Lubricating Intravaginal Ring to Relieve the Symptoms of Vaginal Dryness
Brief Title: Preliminary Study of a Vaginal Lubrication Ring to Treat the Symptoms of Vaginal Dryness
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: J3 Bioscience, Inc. (Industry)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 67709
Record Dates: First submitted 2014-01-03; First posted 2014-01-07 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Menopausal and Perimenopausal Disorder, Unspecified; Atrophic Vaginitis
Keywords: Vaginal dryness; Vaginal lubrication; Post-menopausal symptoms; Peri-menopausal symptoms; Urogenital atrophy; Dyspareunia; Painful intercourse
MeSH Terms: conditions — Atrophic Vaginitis; Dyspareunia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Study (Other): Vaginal Lubrication Ring for Vaginal Dryness
  Interventions: Device: Vaginal Lubrication Ring for Vaginal Dryness

INTERVENTIONS:
Device: Vaginal Lubrication Ring for Vaginal Dryness — Participants will be asked to complete 4 study visits and one final follow-up phone call. Each study visit will include a brief vaginal exam where vaginal fluid levels and pH levels are checked and questionnaires are completed. Daily diaries will be completed at home and returned to the study staff at subsequent visits.
  Participants will self-insert the Intravaginal ring on the 1st study visit. The 2nd study visit will occur 3-4 days later.
  The 3rd study visit will occur approximately 7 days after the 1st visit. Participants will remove the device and self-insert a new intravaginal ring.
  The 4th study visit will occur approximately 14 days after the first visit. Participants will remove the intravaginal ring and undergo a final vaginal exam.
  Participants will be called approximately 7 days after the last visit and will be asked about their current vaginal dryness symptoms and how they felt about the device during the study.
  Other Names: VR101; Intravaginal Ring

SUMMARY:
This is a pilot study, assessing the ability and safety of the use of VR101 intravaginal ring to relieve the symptoms of vaginal dryness, in peri and post-menopausal women. VR1010 is designed to release glycerol. The study will assess the duration of lubrication/ moisturization of the vagina with the VR101 intravaginal ring in place (up to 7 days) and participant satisfaction of the device.

Study participants will insert the intravaginal ring and leave it in place for an initial 7 days and then repeat this process a 2nd time. Participants will respond to questionnaires, complete a daily diary and come in for 4 separate study visits. Each study visit will involve a brief vaginal exam.

Upon removal of the initially inserted device (7 days after first study visit), participants will insert a second device for an additional 7 days and undergo the same evaluation.

DETAILED DESCRIPTION:
Vaginal dryness affects many women, although they frequently do not bring up the topic with their doctors. Vaginal dryness can dramatically affect women's lifestyle, in particular their sexual activity and relationship with their partner. Since we believe that living with uncomfortable vaginal dryness does not have to be part of aging, we intend to conduct this study to evaluate a lubricating vaginal ring developed to ease symptoms caused by vaginal dryness.

The objectives of this study are to obtain preliminary data on the ability of the VR101 intravaginal ring to relieve the symptoms of vaginal dryness in peri- and post-menopausal women. Effectiveness will be measured in two ways:

1. Vaginal health index scoring assessed by a member of the research team
2. Participant answers to questionnaires

Study objectives will assess the following:

1. Successful placement of VR101 intravaginal ring into the vagina
2. Ease of insertion and removal
3. Comfort and fit
4. Lubrication/ moisturization of the vagina

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Females over 35 years of age at the time of enrollment
* Willing to comply with study visit schedule
* Self-reported peri- or post-menopausal women with self-reported vaginal dryness
* Willing to abstain from vaginal intercourse while in the study

Exclusion Criteria:

* Use of hormone therapy
* Undergoing any vulvar or vaginal procedures (biopsies, radiation in the last 3 months)
* Active vulvar or vaginal injections/lesions or complaints, as well as undiagnosed abnormal genital bleeding
* History of chronic pelvic pain, interstitial cystitis, vulvar vestibulitis, pelvic inflammatory disease within the past 12 weeks
* Known current clinically evident cervical or vaginal infection
* Postpartum or post-abortion endometritis, unless symptoms resolved at least 12 weeks prior to study entry
* Current persistent, abnormal vaginal bleeding
* History of inability to place an IVR
* History of any abnormality of the vagina resulting in distortion of the vaginal canal or incompatible with IVR placement
* Body habitus, or history of lower genital tract abnormalities or prior surgeries, which may not allow the vagina to be appropriately accessed
* Known or suspected allergy or hypersensitivity to polyurethane or glycerol
* Known current alcohol or illicit drug abuse
* Participants who have not recovered from adverse events due to chemotherapy or radiation treatment for cancer
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any condition that, in the opinion of the investigator or study staff that would constitute contraindications to participation in the study or would compromise ability to comply with the study protocol

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Vaginal lubrication/moisturization | 14 days
  Assessment of patient reported vaginal lubrication/moisturization while the intravaginal ring is inserted.

SECONDARY OUTCOMES:
Comfort and fit of intravaginal ring | 14 days
  Assessment of patient satisfaction with the comfort and fit of the intravaginal ring during the study period.

OTHER OUTCOMES:
Successful vaginal placement and removal | 14 days
  Assessment of patient ability to self-insert and self-remove the intravaginal ring at the initial study visit as well as throughout the 14 day time period of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Margit Janat-Amsbury, MD, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palacios S. Managing urogenital atrophy. Maturitas. 2009 Aug 20;63(4):315-8. doi: 10.1016/j.maturitas.2009.04.009. Epub 2009 Jun 2. PMID 19493638
- [Background] Vaginal atrophy. Managing vaginal dryness and irritation. Mayo Clin Health Lett. 2012 Oct;30(10):6. No abstract available. PMID 23133861
- [Background] Woods NF. An overview of chronic vaginal atrophy and options for symptom management. Nurs Womens Health. 2012 Dec;16(6):482-93; quiz 494. doi: 10.1111/j.1751-486X.2012.01776.x. PMID 23253575
- [Background] Andelloux M. Products for sexual lubrication: understanding and addressing options with your patients. Nurs Womens Health. 2011 Jun-Jul;15(3):253-7. doi: 10.1111/j.1751-486X.2011.01642.x. No abstract available. PMID 21672177
- [Background] Bond S, Horton LS. Management of postmenopausal vaginal symptoms in women. J Gerontol Nurs. 2010 Jul;36(7):3-7. doi: 10.3928/00989134-20100527-96. Epub 2010 Jul 8. PMID 20608584